CLINICAL TRIAL: NCT06252714
Title: Impact of Defecation Posture on Ease of Bowel Movements in Patients With a Rectocele.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-090
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Pelvic Organ Prolapse; Rectocele; Bowel Dysfunction
Keywords: defecation posture modification device; defecation posture
MeSH Terms: conditions — Pelvic Organ Prolapse; Rectocele; Intestinal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Defecation Posture Modification Device (Experimental): Patients will be given a Squatty Potty Device
  Interventions: Device: Defecation Posture Modification Device

INTERVENTIONS:
Device: Defecation Posture Modification Device — Patients will be asked to use the defecation posture modification device with each bowel movement for two weeks.
  Other Names: Squatty potty

SUMMARY:
The study aims to determine if defecation posture, when using a defecation posture modification device (DPMD), will improve ease of bowel movements in patients with pelvic organ prolapse, specifically rectoceles.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pelvic organ prolapse, including a rectocele (posterior compartment measurements to Stage 2 or greater) that endorse bowel dysfunction, based on our office standard screening questionnaires

Exclusion Criteria:

* Anyone currently using a defecation posture modification device Unwillingness or unable to participate in the study Planned travel, inability to use device during the study period Patient preparing to undergo pelvic reconstructive surgery prior to the end of the study period Presence of ileostomy/colostomy Bowel disease such as Crohn's disease or Ulcerative Colitis Daily opiate use Wheelchair bound If device may pose fall or safety hazard risk to patient, such as need for walker or cane for ambulation.

Patients weighing over 250 lbs, per manufacturer guidelines for the device Inability to understand English Pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Straining with bowel movements | 2 weeks
  Patients will assess straining with bowel movement on a 0 -10 numeric scale. The scale is called straining or ease with bowel movements. The number 0 indicates no straining and the number 10 indicates maximal straining with bowel movement.

SECONDARY OUTCOMES:
Colorectal-Anal Distress Inventory 8 | 2 weeks
  validated questionnaire to assess bowel function. The colorectal-anal distress inventory 8 is a validated questionnaire that asks 8 questions regarding bowel movements. The question is a YES or NO question. If they respond with YES, they respond with how bothersome they symptoms are. The scale is 1-4 with the number 1 being not at all bothersome and the number 4 being quite a bit bothersome.
Consistency of stool | 2 weeks
  Bristol stool scale will be used to describe stool consistency. The Bristol stool scale is rated on Type 1- Type 7 describing the consistency of stool. Type 1 is hard lumps ranging to Type 7 which describes entirely watery and liquid stool. The patient is provided with a visual scale to help assist in answering the questions.
Use of laxative medication | 2 weeks
  patients will log any laxative medication used
Ease of device use | 2 weeks
  patients will be asked questions regarding satisfaction with and ease of use of device. When asked regarding satisfaction of the device they are asked on an 11 point numeric scale with 0 being not satisfied and 10 being very satisfied.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Cincinnati Urogynecology Associates, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No